CLINICAL TRIAL: NCT05239195
Title: DirEct Versus VIdeo LaryngosCopE Trial
Acronym: DEVICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Jonathan Casey, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 211272
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Acute Respiratory Failure
Keywords: Critical Illness; Emergency Airway Management; Tracheal intubation; Video laryngoscope; Direct laryngoscope
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Laryngoscope Group (Active Comparator): For patients assigned to the video laryngoscope group, the operator will use a video laryngoscope on the first laryngoscopy attempt. A video laryngoscope will be defined as a laryngoscope with a camera and a video screen. Trial protocol will not dictate the brand of video laryngoscope.
  Interventions: Other: Video Laryngoscope
- Direct Laryngoscope Group (Active Comparator): For patients assigned to the direct laryngoscope group, the operator will use a direct laryngoscope on the first laryngoscopy attempt. A direct laryngoscope will be defined as a laryngoscope without a camera or a video screen. Trial protocol will not dictate the brand of direct laryngoscope or the blade shape.
  Interventions: Other: Direct Laryngoscope

INTERVENTIONS:
Other: Video Laryngoscope — Laryngoscope with a camera and a video screen
  Arms: Video Laryngoscope Group
Other: Direct Laryngoscope — Laryngoscope without a camera or a video screen
  Arms: Direct Laryngoscope Group

SUMMARY:
Clinicians perform rapid sequence induction, laryngoscopy, and tracheal intubation for more than 5 million critically ill adults as a part of clinical care each year in the United States. Failure to intubate the trachea on the first attempt occurs in more than 10% of all tracheal intubation procedures performed in the emergency department (ED) and intensive care unit (ICU). Improving clinicians rate of intubation on the first attempt could reduce the risk of serious procedural complications.

In current clinical practice, two classes of laryngoscopes are commonly used to help clinicians view the larynx while intubating the trachea: a video laryngoscope (equipped with a camera and a video screen) and a direct laryngoscope (not equipped with a camera or video screen). For nearly all laryngoscopy and intubation procedures performed in current clinical practice, clinicians use either a video or a direct laryngoscope. Prior research has shown that use of a video laryngoscope improves the operator's view of the larynx compared to a direct laryngoscope. Whether use of a video laryngoscope increases the likelihood of successful intubation on the first attempt remains uncertain. A better understanding of the comparative effectiveness of these two common, standard-of-care approaches to laryngoscopy and intubation could improve the care clinicians deliver and patient outcomes.

DETAILED DESCRIPTION:
Clinicians frequently perform tracheal intubation of critically ill patients in the emergency department (ED) or intensive care unit (ICU). In 10-20% of emergency tracheal intubations, clinicians are unable to intubate the trachea on the first attempt, which increases the risk of peri-intubation complications. Successful laryngoscopy and tracheal intubation requires using a laryngoscope to [1] visualize the larynx and vocal cords and [2] create a pathway through which an endotracheal tube can be advanced through the oropharynx and larynx and into the trachea.

In current clinical practice, two classes of laryngoscopes are commonly used by clinicians to view the larynx while intubating the trachea: a video laryngoscope (equipped with a camera and a video screen) and a direct laryngoscope (not equipped with a camera or video screen). Clinicians use either a video laryngoscope or a direct laryngoscope as standard of care for every laryngoscopy and intubation procedure performed in current clinical practice.

Direct Laryngoscope: The Macintosh direct laryngoscope consists of a battery-containing handle and a blade with a light source. The operator achieves a direct line of sight -from the operator's eye through the mouth to the larynx and trachea - by using the laryngoscope blade to displace the tongue and elevate the epiglottis.

Video Laryngoscope: Video laryngoscopes consist of a fiberoptic camera and light source near the tip of the laryngoscope blade, which transmits images to a video screen. The position of the camera near the tip of the laryngoscope blade facilitates visualization of the larynx and trachea.

Use of a video laryngoscope and use of a direct laryngoscope are both common, standard-of-care approaches the clinicians use to perform tracheal intubation in the ED and ICU in current clinical care.

Currently, it is unknown whether use of a video laryngoscope or use of a direct laryngoscope has any effect on successful intubation on the first attempt or any other outcome. Some prior research has raised the hypothesis that using a video laryngoscope would increase clinicians' rate of successful intubation on the first attempt by facilitating the view of the larynx. Some prior research has raised the hypothesis that using a direct laryngoscope would increase clinicians' rate of successful intubation on the first attempt by facilitating a clear pathway for placement of the tube through the mouth into the trachea.

To date, 8 small single-center randomized trials and one 371-patient multicenter randomized clinical trial have been conducted under waiver of or alteration of informed consent to compare use of a video vs a direct laryngoscope in the setting of emergency tracheal intubation in the ED or ICU. Two of these trials provide the most direct preliminary data for this proposal. The "Facilitating EndotracheaL intubation by Laryngoscopy technique and apneic Oxygenation Within the ICU (FELLOW)" randomized clinical trial, conducted under waiver of informed consent, compared these two standard-of-care approaches during 150 emergency tracheal intubations at Vanderbilt University Medical Center, finding no difference in the rate of successful intubation on the first attempt between use of a video and use of a direct laryngoscope. The "McGrath Mac Videolaryngoscope Versus Macintosh Laryngoscope for Orotracheal Intubation in the Critical Care Unit (MACMAN)" randomized clinical trial among 371 critically ill adults found no difference between use of a video vs direct laryngoscope in the rate of successful intubation on the first attempt. However, a hypothesis-forming post-hoc exploratory analysis of peri-intubation complications suggested that use of a video laryngoscope may be associated with a higher rate of complications than direct laryngoscope (9.5% vs 2.8%, respectively, p=0.01). These trials were underpowered to rule out small but clinically significant differences in first pass success, and were limited to intubations performed by inexperienced trainees in one practice setting (intensive care units), but they demonstrated hypothesis-generating findings requiring validation in larger trials that reflect the full spectrum of settings, operator specialties, and operator experience levels in which emergency tracheal intubation is routinely performed.

Because of the imperative to optimize emergency tracheal intubation in clinical care, the common use of both video and direct laryngoscopes in current clinical practice, and the lack of definitive data from randomized trials to definitively inform whether use of a video laryngoscope or a direct laryngoscope effects the rate of successful intubation on the first attempt, examining whether one approach increases the odds of successful intubation on the first attempt represents an urgent research priority. To address this knowledge gap, the investigators propose to conduct a large, multicenter, randomized clinical trial comparing use of a video laryngoscope versus use of a direct laryngoscope with regard to successful intubation on the first attempt among critically ill adults undergoing tracheal intubation in the ED or ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patient is located in a participating unit.
* Planned procedure is orotracheal intubation using a laryngoscope.
* Planned operator is a clinician expected to routinely perform tracheal intubation in the participating unit.

Exclusion Criteria:

* Patient is known to be less than 18 years old.
* Patient is known to be pregnant.
* Patient is known to be a prisoner.
* Immediate need for tracheal intubation precludes safe performance of study procedures.
* Operator has determined that use of a video laryngoscope or use of a direct laryngoscope is required or contraindicated for the optimal care of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1420 (Actual)
Dates: Start 2022-03-19 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Semler, MD, MSc, Principal Investigator — Vanderbilt University Medical Center; Adit A Ginde, MD, MPH, Principal Investigator — University of Colorado, Denver; Matthew E Prekker, MD, MPH, Study Chair — Hennepin County Medical Center, Minneapolis; Stacy A Trent, MD, MPH, Study Chair — Denver Health Medical Center; Brian E Driver, MD, Study Chair — Hennepin County Medical Center, Minneapolis; Jonathan D Casey, MD, MSc, Study Director — Vanderbilt University Medical Center
Locations (12):
- United States (12):
  - UAB Hospital, Birmingham, Alabama
  - University of Colorado Denver, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Ochsner Medical Center | Ochsner Health System, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor Scott & White Health, Temple, Texas
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Following publication, individual patient data will be made available for sharing to researchers with 1) a signed data access agreement, 2) research testing a hypothesis, 3) a protocol that has been approved by an institutional review board, and 4) a proposal that has received approval from the principal investigator.
Supporting Information: Study Protocol, SAP
Time Frame: Following publication. No end date
Access Criteria: 1. a signed data access agreement
  2. research testing a hypothesis
  3. a protocol that has been approved by an institutional review board
  4. a proposal that has received approval from the principal investigator

REFERENCES:
- [Derived] Prekker ME, Driver BE, Trent SA, Resnick-Ault D, Seitz KP, Russell DW, Gaillard JP, Latimer AJ, Ghamande SA, Gibbs KW, Vonderhaar DJ, Whitson MR, Barnes CR, Walco JP, Douglas IS, Krishnamoorthy V, Dagan A, Bastman JJ, Lloyd BD, Gandotra S, Goranson JK, Mitchell SH, White HD, Palakshappa JA, Espinera A, Page DB, Joffe A, Hansen SJ, Hughes CG, George T, Herbert JT, Shapiro NI, Schauer SG, Long BJ, Imhoff B, Wang L, Rhoads JP, Womack KN, Janz DR, Self WH, Rice TW, Ginde AA, Casey JD, Semler MW; DEVICE Investigators and the Pragmatic Critical Care Research Group. Video versus Direct Laryngoscopy for Tracheal Intubation of Critically Ill Adults. N Engl J Med. 2023 Aug 3;389(5):418-429. doi: 10.1056/NEJMoa2301601. Epub 2023 Jun 16. PMID 37326325
- [Derived] Prekker ME, Driver BE, Trent SA, Resnick-Ault D, Seitz K, Russell DW, Gandotra S, Gaillard JP, Gibbs KW, Latimer A, Whitson MR, Ghamande S, Vonderhaar DJ, Walco JP, Hansen SJ, Douglas IS, Barnes CR, Krishnamoorthy V, Bastman JJ, Lloyd BD, Robison SW, Palakshappa JA, Mitchell S, Page DB, White HD, Espinera A, Hughes C, Joffe AM, Herbert JT, Schauer SG, Long BJ, Imhoff B, Wang L, Rhoads JP, Womack KN, Janz D, Self WH, Rice TW, Ginde AA, Casey JD, Semler MW; DEVICE investigators and the Pragmatic Critical Care Research Group. DirEct versus VIdeo LaryngosCopE (DEVICE): protocol and statistical analysis plan for a randomised clinical trial in critically ill adults undergoing emergency tracheal intubation. BMJ Open. 2023 Jan 13;13(1):e068978. doi: 10.1136/bmjopen-2022-068978. PMID 36639210

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group
Started | 707 | 713
Completed | 705 | 712
Not Completed | 2 | 1
Not completed — After enrollment, discovered to be a person experiencing incarceration. | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group | Total
Number analyzed (Participants) | 705 | 712 | 1417
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [36 to 66] | 55 [39 to 67] | 55 [38 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 240 | 258 | 498
  Male | 465 | 454 | 919
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race or ethnic group: Non-Hispanic White | 360 | 346 | 706
  Race or ethnic group: Non-Hispanic Black | 166 | 167 | 333
  Race or ethnic group: Hispanic | 101 | 94 | 195
  Race or ethnic group: Other | 61 | 84 | 145
  Race or ethnic group: Not reported | 17 | 21 | 38
Region of Enrollment [Number; unit: participants]
  United States | 705 | 712 | 1417

OUTCOME MEASURES:

1. Primary Outcome: Number of Intubations With Successful Intubation on the First Attempt
Description: The primary outcome is defined as placement of an endotracheal tube in the trachea with a single insertion of a laryngoscope blade into the mouth and EITHER a single insertion of an endotracheal tube into the mouth OR a single insertion of a bougie into the mouth followed by a single insertion of an endotracheal tube over the bougie into the mouth.
Time Frame: Duration of procedure (minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group
Number analyzed (Participants) | 705 | 712
Participants | 600 | 504

2. Secondary Outcome: Number of Participants With Severe Complications of Tracheal Intubation
Description: The secondary outcome is defined as the number of patients who experienced one or more of the following occurring between induction and 2 minutes after successful intubation:
  * Severe hypoxemia (lowest oxygen saturation measured by pulse oximetry < 80%);
  * Severe hypotension (systolic blood pressure < 65 mm Hg or new or increased vasopressor administration);
  * Cardiac arrest not resulting in death within 1 hour of intubation; or
  * Cardiac arrest resulting in death within 1 hour of induction
Time Frame: from induction to 2 minutes following tracheal intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group
Number analyzed (Participants) | 705 | 712
Participants | 151 | 149

3. Other Pre Specified Outcome: Duration of Laryngoscopy and Tracheal Intubation
Description: The interval (in seconds) between the first insertion of a laryngoscope blade into the mouth and the final placement of an endotracheal tube or tracheostomy tube in the trachea.
Time Frame: Duration of procedure (minutes)
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group
Number analyzed (Participants) | 705 | 712
Seconds | 38 [26 to 60] | 46 [30 to 83]

4. Other Pre Specified Outcome: Number of Laryngoscopy Attempts
Time Frame: Duration of procedure (minutes)
Population: A subset of patients were missing this data variable.
Measure: Count of Participants; unit: Participants
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group
Number analyzed (Participants) | 704 | 706
Participants
  Number of times a laryngoscope entered the patient's mouth (reported by observer) - 1 | 636 | 546
  Number of times a laryngoscope entered the patient's mouth (reported by observer) - 2 | 54 | 127
  Number of times a laryngoscope entered the patient's mouth (reported by observer) - 3+ | 14 | 33

5. Other Pre Specified Outcome: Number of Attempts to Cannulate the Trachea With a Bougie or an Endotracheal Tube
Time Frame: Duration of procedure (minutes)
Population: Data was not available for entire patient population.
Measure: Number; unit: number of events
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group
Number analyzed (Participants) | 705 | 707
number of events
  Endotracheal Tube - 1: number analyzed (Participants) | 704 | 705
  Endotracheal Tube - 1 | 646 | 620
  Endotracheal Tube - 2: number analyzed (Participants) | 704 | 705
  Endotracheal Tube - 2 | 43 | 66
  Endotracheal Tube - 3+: number analyzed (Participants) | 704 | 705
  Endotracheal Tube - 3+ | 15 | 19
  Bougie - 0 | 364 | 330
  Bougie - 1 | 316 | 317
  Bougie - 2 | 19 | 33
  Bougie - 3+ | 6 | 27

6. Other Pre Specified Outcome: Successful Intubation on the First Attempt Without a Severe Complication
Description: This outcome reports the number of participants that experienced successful intubation on the first attempt without experiencing complications, a composite of two independent outcomes: successful intubation on the first attempt (the primary outcome of the trial) and severe complication (the secondary outcome of the trial).
Time Frame: from induction to 2 minutes following tracheal intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group
Number analyzed (Participants) | 705 | 712
Participants | 484 | 420

7. Other Pre Specified Outcome: Reason for Failure to Intubate on the First Attempt
Description: Providers could give more than one reason for failure to intubate on the first attempt for each intubation (not mutually exclusive). In addition, data on the reason for failure to intubate on the first attempt was missing for 23 patients in the video laryngoscope group and 40 patients in the direct laryngoscope group.
  Reason for failure among those who did not meet the primary outcome (successful intubation on the first attempt):
  * Inadequate view of the larynx
  * Inability to intubate the trachea with an endotracheal tube
  * Inability to cannulate the trachea with a bougie
  * Attempt aborted due to change in patient condition (e.g., worsening hypoxemia, hypotension, bradycardia, vomiting, bleeding)
  * Technical failure of the laryngoscope (e.g., battery, light source, camera, screen)
  * Other
  * Not Reported
Time Frame: Duration of procedure (minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group
Number analyzed (Participants) | 705 | 712
Participants
  Inadequate view of the larynx | 26 | 123
  Inability to intubate the trachea with an endotracheal tube | 44 | 32
  Inability to cannulate the trachea with a bougie | 7 | 19
  Attempt aborted due to change in patient condition | 2 | 14
  Technical failure of the laryngoscope (e.g., battery, light source, camera, screen) | 2 | 4
  Other | 13 | 10
  Not Reported | 23 | 40

8. Other Pre Specified Outcome: Operator-reported Aspiration
Time Frame: from induction to 2 minutes following tracheal intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group
Number analyzed (Participants) | 705 | 712
Participants | 7 | 12

9. Other Pre Specified Outcome: Esophageal Intubation
Time Frame: from induction to 2 minutes following tracheal intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group
Number analyzed (Participants) | 705 | 712
Participants | 6 | 9

10. Other Pre Specified Outcome: Injury to the Teeth
Time Frame: from induction to 2 minutes following tracheal intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group
Number analyzed (Participants) | 705 | 712
Participants | 3 | 2

11. Other Pre Specified Outcome: ICU-free Days in the First 28 Days
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group
Number analyzed (Participants) | 705 | 712
days | 20 [0 to 25] | 19 [0 to 24]

12. Other Pre Specified Outcome: Ventilator Free Days in the First 28 Days
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group
Number analyzed (Participants) | 705 | 712
days | 24 [0 to 26] | 23 [0 to 26]

13. Other Pre Specified Outcome: All-cause In-hospital Mortality
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group
Number analyzed (Participants) | 705 | 712
Participants | 184 | 191

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Video Laryngoscope Group | Direct Laryngoscope Group
All-Cause Mortality (participants affected / at risk) | 184/705 | 191/712
Serious Adverse Events (participants affected / at risk) | 0/705 | 0/712
Other Adverse Events (participants affected / at risk) | 0/705 | 0/712

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT05239195/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT05239195/SAP_001.pdf